CLINICAL TRIAL: NCT06490588
Title: The Use of Sevoflurane to Test the Concept of Intra-individual Variability in Bispectral Index Monitor and Cognitive Reserve by Examining Time to Emergence and Recovery
Brief Title: Use of Sevoflurane to Test Concept of Cognitive Reserve
Status: Not yet recruiting | Type: Observational
Sponsor: Los Angeles General Medical Center (Other)
Responsible Party: Principal Investigator, Jody Chou, Physician Specialist, Los Angeles General Medical Center
Other Study IDs: HS-22-00653
Record Dates: First submitted 2024-06-25; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Cognitive Reserve; BIS
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sevoflurane — No intervention

SUMMARY:
Previous pilot study had demonstrated a correlation between cognitive reserve and BIS variability during steady state of anesthesia. This study, we intend to evaluate the association between BIS variability and emergence and recovery time from anesthesia.

DETAILED DESCRIPTION:
Cognitive reserve (CR) refers to an individual's ability to resist damage to the brain and is thought to be associated with an individual's education, cognitive stimulation, and physical activity. Those with greater CR have protection against degenerative brain changes such as dementia. Currently, CR is evaluated through a host of proxy tests such as questionnaires aimed to assess various aspects of cognitive function. These ways of measuring CR test directly only on an individual's ability to perform certain tasks when the brain is in its "unchallenged" state. However, this approach poses significant limitations since CR is developed as a concept representing the physiological brain reserve that helps counter the clinical manifestation of a diseased or "challenged" brain. A method that simulates a state of "challenged" brain during CR measurement may provide a more precise assessment of CR.

Anesthetic agents are known to reversibly alter brain function resulting in a state of sedation or amnesia. Whether this way of brain "challenge" can provide information on CR is unknown.

A previous study showed preliminary evidence that patients with higher CR correlates with less variability in bispectral index (BIS) during steady state of anesthesia with inhaled anesthetic sevoflurane (1). While the result of this study is encouraging, further study is needed to develop the concept of using anesthetic agents to evaluate CR. Specifically, a study investigating the correlation between intraoperative BIS variability and timing of clinical recovery from anesthesia will be necessary. This will further elucidate how to use anesthetic agent for the evaluation of CR.

Building on the previous study result and the concept that higher CR means higher resilience against brain function in a "challenged" state, we hypothesize that less intraoperative BIS variability correlates with shorter recovery time from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* - Minimal completion of high-school education
* Adult patient < 85 years of age
* No prior known history of cognitive/brain disease
* ASA class I-II
* Undergoing general anesthesia with sevoflurane for maintenance anesthesia
* Same-day surgery
* Elective procedures
* No prior history of cardiac disease

Exclusion Criteria:

* - History of chronic pain
* Perioperative use of anesthetic agents other than propofol, fentanyl, dilaudid, and sevoflurane
* History of alcohol/substance druge abuse
* Psychiatric history
* Morbid history
* History of OSA, stroke, or TIA
* Blindness
* Deafness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I or II
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
intraoperative BIS variability | 360 minutes

SECONDARY OUTCOMES:
time to recovery | 120 minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernaiz Alonso C, Tanner JJ, Wiggins ME, Sinha P, Parvataneni HK, Ding M, Seubert CN, Rice MJ, Garvan CW, Price CC. Proof of principle: Preoperative cognitive reserve and brain integrity predicts intra-individual variability in processed EEG (Bispectral Index Monitor) during general anesthesia. PLoS One. 2019 May 23;14(5):e0216209. doi: 10.1371/journal.pone.0216209. eCollection 2019. PMID 31120896